CLINICAL TRIAL: NCT03232814
Title: Walk on: A Community-based Approach to Promote Participation in Physical Activity Among Men Treated for Colorectal Cancer
Brief Title: Walk on: A Community-based Approach to Increase Physical Activity Among Men Treated for Colorectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were recruited due to a lack of referrals.
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, Associate Professor, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WBCP:PA/CR
Record Dates: First submitted 2017-07-23; First posted 2017-07-28 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-based walking (Experimental): Participants will engage in one supervised outdoor group-based walking session per week for the 8 week program.
  Interventions: Behavioral: Group-based walking

INTERVENTIONS:
Behavioral: Group-based walking — The walking prescription will be progressive in nature. The program will begin with participants walking for approximately 20 minutes in weeks 1-3. This will gradually increase to approximately 30 minutes in weeks 4-6. Finally, this will increase to 45-60 minutes in weeks 7-8. The program will promote walking at a moderate intensity as assessed by Borg's Rating of Perceived Exertion scale. Each session will be preceded by a brief warm-up and followed by a brief cool-down period.

SUMMARY:
In Canada, over 102,900 men are diagnosed with cancer each year. Of these, 81,000 are diagnosed with colorectal cancer and an estimated 65% are expected to survive the disease for at least 5 years. Men who have completed treatment for colorectal cancer face many adverse physical, cognitive, psychological, and social effects. The Wellness Beyond Cancer Program at The Ottawa Hospital is a cancer survivorship program that helps people who have completed treatment for cancer, including men diagnosed with colorectal cancer, manage these effects. The Wellness Beyond Cancer Program does this through education and referral to supportive care services and programs offered throughout the city of Ottawa.

Group-based physical activity programs are one of the varied services and programs available to adults diagnosed with cancer in Ottawa. Such programs are offered through the Ottawa Regional Cancer Foundation (http://www.ottawacancer.ca) and Breast Cancer Action Ottawa (http://bcaott.ca). Research on these programs show that group-based physical activity can improve disease and treatment-related effects while promoting overall quality of life amongst women with cancer. However, few of these programs have targeted men, even though their needs and preferences have been shown to be very different from women. While men diagnosed with colorectal cancer might also benefit from group-based physical activity programs offered in the community, it is not known if such programs would effectively reach them and what the impact would be on their quality of life after cancer treatment.

It is believed that a men's group-based walking program could be an effective way to reach men and promote quality of life after cancer treatment. Therefore, a sustainable 8-week group-based walking program was developed. This project will seek to explore the feasibility and potential benefits of the program among men who have completed treatment for colorectal cancer and who are referred to the program from staff at the Wellness Beyond Cancer Program in a prospective single-arm trial.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 years of age or older;
2. Have completed treatment for colorectal cancer <1 year;
3. Willing to provide informed consent to participate in this study and willing to follow the study protocol;
4. Have the ability to walk without the use of an assistive device (including a cane) or the help of another person;
5. Able to read and understand English;
6. Medically cleared to participate in the walking program as determined by their referring Wellness Beyond Cancer Program healthcare provider.

Exclusion Criteria:

1. Congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, uncontrolled angina, uncontrolled arrhythmia, myocardial infarction, major heart surgery, stroke, or pulmonary embolus;
2. Uncontrolled hypertension (systolic blood pressure>200 mm Hg and/or diastolic blood pressure >110 mm Hg);
3. The use of supplemental oxygen;
4. Severe arthritis (i.e., osteoarthritis or rheumatoid arthritis);
5. History of chest pain or severe shortness of breath either at rest or when engaging in physical activity;
6. Hip fracture, hip or knee replacement in the past 6 months;
7. Currently enrolled in another study involving a physical activity intervention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | Through study completion, an average of 8 weeks
  The number of men who enrol in the study out of the number who are referred.
Retention rates | Through study completion, an average of 8 weeks
  The number of men who complete the intervention and all scheduled assessments.
Adherence rates | Through study completion, an average of 8 weeks
  The number of walking sessions men engage in out of the total recommended as part of the intervention.

SECONDARY OUTCOMES:
Change in Physical Activity Behaviour: Leisure Time Exercise Questionnaire (Godin & Shephard, 1985) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported physical activity (over the past 7 days) from baseline to post-intervention.
Change in Quality of Life: Functional Assessment of Cancer Therapy (FACT)-Colorectal (Ward et al., 1999; Yost et al. 2005) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported quality of life from baseline to post-intervention.
Change in Cognitive Functioning: FACT-Cognitive Function (Wagner et al., 2004) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported cognitive functioning from baseline to post-intervention.
Change in Affect: Positive and Negative Affect Schedule (Watson et al., 1988) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported affect from baseline to post-intervention.
Change in Depression: Center for Epidemiologic Studies Depression Scale 10-item Revised (Eaton et al., 2004; Radloff, 1977) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported depressive symptoms from baseline to post-intervention.
Change in Social Support: Relatedness to Others in Physical Activity Scale (Wilson & Bengoechea, 2010) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported perceptions of social support from baseline to post-intervention.
Change in Physical Self-Perceptions: Physical Self Description Questionnaire Short-Form (Marsh et al., 2010) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported physical competence, confidence, and self-esteem from baseline to post-intervention.
Change in Stress: Perceived Stress Scale (Cohen et al., 1982) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported perceptions of stress from baseline to post-intervention.
Change in Fatigue: Functional Assessment of Chronic Illness Therapy-Fatigue Scale (Yellen et al., 1997) | Baseline (week 0) and post-intervention (week 8)
  Change in participants' self-reported perceptions of fatigue from baseline to post-intervention.
Participants' Overall Experiences: Qualitative Interviews | Post-intervention (week 8)
  Participants' perspectives on how the intervention contributed to their behavioural, physical, psychological and social functioning, as well as their overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brunet, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Eaton WW, Muntaner C, Smith C, Tien A, Ybarra M. Center for Epidemiologic Studies Depression Scale: Review and revision (CESD and CESD-R), in The Use of Psychological Testing for Treatment Planning and Outcomes Assessment, M.E. Maruish, Editor. 2004, Lawrence Erlbaum: Mahwah, NJ. p. 363-377.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Marsh HW, Martin AJ, Jackson S. Introducing a short version of the physical self description questionnaire: new strategies, short-form evaluative criteria, and applications of factor analyses. J Sport Exerc Psychol. 2010 Aug;32(4):438-82. doi: 10.1123/jsep.32.4.438. PMID 20733208
- [Background] Radloff LS. The CES-D scale: a self-report depression scale for research in the general population. Applied Psychological Measurement, 1977. 1: p. 385-401.
- [Background] Wagner L, Lai J-S, Cella D, Sweet J, Forrestal S. Chemotherapy-related cognitive deficits: development of the FACT-Cog instrument. Ann Behav Med, 2004. 27: p. S10.
- [Background] Ward WL, Hahn EA, Mo F, Hernandez L, Tulsky DS, Cella D. Reliability and validity of the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) quality of life instrument. Qual Life Res. 1999 May;8(3):181-95. doi: 10.1023/a:1008821826499. PMID 10472150
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Wilson PM, Bengoechea EG. The relatedness to others in physical activity scale: evidence for structural and criterion validity. Journal of Applied Biobehavioral Research, 2010. 15(2): p. 61-87.
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Yost KJ, Cella D, Chawla A, Holmgren E, Eton DT, Ayanian JZ, West DW. Minimally important differences were estimated for the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) instrument using a combination of distribution- and anchor-based approaches. J Clin Epidemiol. 2005 Dec;58(12):1241-51. doi: 10.1016/j.jclinepi.2005.07.008. Epub 2005 Oct 13. PMID 16291468